CLINICAL TRIAL: NCT04255225
Title: Making Activity Time for Cognitive Health (MATCH)
Brief Title: Making Activity Time for Cognitive Health
Acronym: MATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Edward McAuley, Shahid and Ann Carlson Khan Professor in Applied Health Sciences, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UIUC_IRB_16912
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer; Cancer-related Problem/Condition; Cognitive Impairment; Physical Activity
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction; Motor Activity | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 10-minute Treadmill Walking (Experimental): All participants will walk on the treadmill and perform a battery of cognitive tasks immediately prior and immediately after the walking session. Participants will be randomized the length of time spent walking on the treadmill: 10, 20 or 30 minutes.
  Interventions: Behavioral: Walking for 10 minutes
- 20-minute Treadmill Walking (Experimental): All participants will walk on the treadmill and perform a battery of cognitive tasks immediately prior and immediately after the walking session. Participants will be randomized the length of time spent walking on the treadmill: 10, 20 or 30 minutes.
  Interventions: Behavioral: Walking for 20 minutes
- 30-minute Treadmill Walking (Experimental): All participants will walk on the treadmill and perform a battery of cognitive tasks immediately prior and immediately after the walking session. Participants will be randomized the length of time spent walking on the treadmill: 10, 20 or 30 minutes.
  Interventions: Behavioral: Walking for 30 minutes

INTERVENTIONS:
Behavioral: Walking for 10 minutes — Participants will walk on a treadmill for 10 minutes at a moderate intensity.
  Arms: 10-minute Treadmill Walking
Behavioral: Walking for 20 minutes — Participants will walk on a treadmill for 20 minutes at a moderate intensity.
  Arms: 20-minute Treadmill Walking
Behavioral: Walking for 30 minutes — Participants will walk on a treadmill for 30 minutes at a moderate intensity.
  Arms: 30-minute Treadmill Walking

SUMMARY:
Approximately 75% of cancer survivors experience some degree of cognitive deficit throughout their cancer experience, with upwards of one third of breast cancer survivors reporting impairments up to a decade after treatment. Chemotherapy and adjuvant therapy to remove cancerous tissue can result in deficits in attention, speed of processing, memory, and quality of life. Physical activity has been associated with a number of health benefits for breast cancer survivors including improvements in cognitive function. The investigators recently reported on the beneficial effects of acute exercise, or single sessions of physical activity, on processing speed and spatial working memory in breast cancer survivors, suggesting that acute bouts of physical activity may mitigate select domains of CRCI. Specifically, survivors in this study demonstrated faster processing speed, and trended towards faster and more accurate spatial working memory, after thirty minutes of moderate-intensity walking compared to seated rest. But half an hour of walking may be challenging to certain subgroups of survivors, particularly those who are deconditioned or with significant barriers to longer walks. With a renewed focus on un-bouted physical activity and avoiding inactivity during survivorship, it is important to better understand the dose or volume of exercise responsible for providing breast cancer survivors with the greatest cognitive benefits. The investigators examined the effects of varying durations of exercise (e.g., 10, 20 and 30 minutes) on cognitive function in breast cancer survivors to identify the optimal length of acute exercise. Findings from this study will inform new guidelines for acute exercise after cancer.

ELIGIBILITY:
Inclusion Criteria:

* women over the age of 18
* diagnosis of breast cancer
* no longer undergoing treatment
* fluent in English
* no history of dementia or organic brain syndrome
* not currently pregnant
* able to walk unassisted
* no health reasons that would prevent ability to exercise
* not currently enrolled in another exercise research study
* reported trouble with memory/concentration
* physician's consent

Exclusion Criteria:

* male
* no diagnosis of breast cancer
* under 18 years of age
* currently undergoing treatment for breast cancer
* inability to communicate in English
* history of dementia or organic brain syndrome
* pregnant
* unable to walk unassisted
* other health reasons that may prevent ability to exercise
* enrolled in another exercise research study
* no reported trouble with memory or concentration
* non-consent of physician

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants will be female breast cancer survivors.
Enrollment: 50 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in working memory by walking as a function of walking duration (10, 20 or 30 minutes) | 1 year
  All participants will complete both a walking and a sitting session, but the duration of these sessions will be determined randomly. Prior to each session, participants will complete a cognitive battery consisting of a working memory task (Spatial Working Memory domain). They will then complete the same cognitive battery immediately after the session. Accuracy ranges from 0-100% and reaction time ranges from 0-5000 milliseconds.
Change in attention by walking as a function of walking duration (10, 20 or 30 minutes) | 1 year
  All participants will complete both a walking and a sitting session, but the duration of these sessions will be determined randomly. Prior to each session, participants will complete a cognitive battery consisting of an attention task (Flanker task). They will then complete the same cognitive battery immediately after the session. Accuracy ranges from 0-100% and reaction time ranges from 0-5000 milliseconds.
Change in cognitive flexibility by walking as a function of walking duration (10, 20 or 30 minutes) | 1 year
  All participants will complete both a walking and a sitting session, but the duration of these sessions will be determined randomly. Prior to each session, participants will complete a cognitive battery consisting of a cognitive flexibility task (Task Switching Paradigm). They will then complete the same cognitive battery immediately after the session. Accuracy ranges from 0-100% and reaction time ranges from 0-5000 milliseconds.
Change in processing speed by walking as a function of walking duration (10, 20 or 30 minutes) | 1 year
  All participants will complete both a walking and a sitting session, but the duration of these sessions will be determined randomly. Prior to each session, participants will complete a cognitive battery consisting of a processing speed task (Letter Comparison task). They will then complete the same cognitive battery immediately after the session. Accuracy ranges from 0-100% and reaction time ranges from 0-5000 milliseconds.

SECONDARY OUTCOMES:
Lifestyle physical activity as a predictor of change in cognitive function (executive function domains: working memory, attention/inhibition/cognitive flexibility and processing speed) after acute exercise | 1 year
  Investigators are interested in determining what lifestyle factors are associated with significant change in cognition (processing speed, working memory, attention/inhibition, cognitive flexibility) from pre- to post-acute exercise. Lifestyle physical activity will be measured via accelerometer in units of average minutes per day. Higher values indicate greater levels of lifestyle physical activity.
Mental health as a predictor of change in cognitive function (executive function domains: working memory, attention/inhibition/cognitive flexibility and processing speed) after acute exercise | 1 year
  Investigators are interested in determining what mental health factors are associated with significant change in cognition (processing speed, working memory, attention/inhibition, cognitive flexibility) from pre- to post-acute exercise. Mental health factors of interest are anxiety and depression as measured via the Hospital Anxiety and Depression Scale (HADS) questionnaire. Scores range from 0-21 with higher scores indicating increased anxiety and depression.
Body mass index as a predictor of change in cognitive function (executive function domains: working memory, attention/inhibition/cognitive flexibility and processing speed) after acute exercise | 1 year
  Investigators are interested in determining is body mass index associated with significant change in cognition (processing speed, working memory, attention/inhibition, cognitive flexibility) from pre- to post-acute exercise. Body mass index will be measured using the standard kilograms/meters^2. Increased body mass index indicates worsened health.
Change from baseline in anxiety levels after one bout of exercise as assessed by the Hospital Anxiety and Depression Scale (HADS) questionnaire. | 30 minutes
  Participants will complete a short anxiety questionnaire before and after a 30 minute bout of aerobic exercise. The investigators will then compare the pre- and post- values to examine if any changes are present. Scores on the HADS range from 0-21 with higher scores indicating increased anxiety and depression.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salerno EA, Rowland K, Hillman CH, Trinh L, Kramer AF, McAuley E. Dose-Response Effects of Acute Aerobic Exercise Duration on Cognitive Function in Patients With Breast Cancer: A Randomized Crossover Trial. Front Psychol. 2020 Jul 14;11:1500. doi: 10.3389/fpsyg.2020.01500. eCollection 2020. PMID 32760319